CLINICAL TRIAL: NCT07370688
Title: Iron Infusion in Patients Undergoing Transcatheter Aortic Valve Implantation: Study Protocol of the Randomized Controlled IRON-TAVI Trial
Brief Title: Iron Infusion in Patients Undergoing Transcatheter Aortic Valve Implantation
Acronym: IRON TAVI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Rutger-Jan Nuis, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2024-0152
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Aortic Valve Stenosis; Iron Deficiency; TAVI(Transcatheter Aortic Valve Implantation); Cardiovascular Diseases
Keywords: Health-related Quality of Life; Six-Minute Walk Test; Randomized Controlled Trial; Aortic Valve Stenosis; Intravenous Iron Therapy; Kansas City Cardiomyopathy Questionnaire; Functional Recovery; Iron Deficiency; Cardiovascular Diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Iron Deficiencies; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Receiving intravenous iron therapy (ferric carboxymaltose) after TAVI, administered in 1-3 settings over the course of 12 weeks.
  Interventions: Drug: Intravenous ferric carboxymaltose
- Control arm (No Intervention): Receiving standard of care, i.e. no intravenous iron therapy (ferric carboxymaltose) after TAVI.

INTERVENTIONS:
Drug: Intravenous ferric carboxymaltose — The intervention involves the administration of intravenous ferric carboxymaltose (FCM) to correct iron deficiency (ID) in patients with severe aortic stenosis. FCM will be delivered in 1 to 3 settings, depending on the patient's baseline hemoglobin level, body weight, and persistence of ID after the initial administration(s):
  1. Setting-1: After successful TAVI and before hospital discharge, a maximum of 1000 milligrams of FCM will be administered.
  2. Setting-2: A second dose of 500-1000 milligrams FCM will be administered during outpatient-clinic visit if the cumulative iron dosage has not yet been met.
  3. Setting-3: A third dose of 500 milligrams of FCM will be administered at week 12 if ID recurs or persists during follow-up.
  Each dose will be infused using peripheral venous access over at least 15 minutes. The total duration of the intervention is 12 weeks, after which an endpoint outpatient follow-up assessment takes place at week 24 post-TAVI.
  Arms: Intervention arm

SUMMARY:
The aim of the open-label, randomized controlled superiority IRON TAVI trial is to investigate whether intravenous iron therapy (ferric carboxymaltose) improves Health-Related Quality of Life (HRQOL) in patients with severe aortic stenosis (AS) and iron deficiency (ID), undergoing transcatheter aortic valve implantation (TAVI).

The main questions it aims to answer are:

1. Does intravenous iron therapy improve HRQOL after TAVI in patients with severe AS and ID compared to no intravenous iron therapy (standard of care)?
2. Can intravenous iron therapy enhance exercise capacity, as measured by the 6-minute walk test, after TAVI in patients with severe AS and ID compared to no intravenous iron therapy (standard of care)?

The intervention group (receiving iron therapy after TAVI) will be compared to the control group (receiving no iron therapy after TAVI (standard of care)).

Participants will:

* Provide written informed consent
* Be randomly assigned to one of two groups:

  1. Intervention group: receiving intravenous iron therapy after TAVI (1-3 administrations in the course of 12 weeks)
  2. Control group: receiving standard of care (= no iron therapy)
* Complete assessments of HRQOL and the 6-minute walk test at baseline and week 24 after TAVI.
* During follow-up visits, other clinical parameters will be collected (i.e. laboratory status, mortality status, adverse clinical events)

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 65 years
* Patients with severe AS and ID undergoing successful TAVI
* ID defined as Ferritin < 100 ug/L and/or Transferrin saturation < 20%
* Ability to perform assessment of QoL (questionnaire assessment) and EC (6-MWT)
* Signed Informed Consent

Exclusion Criteria:

* Contra-indication for TAVI
* Ferritin > 400 ug/L
* Hemoglobin <5.6 mmol/L or <9 g/dL
* Hemoglobin >8.7 mmol/L or >14 g/dL in men and >8.1 mmol/L or >13 g/dL in women
* Anaemia due to known reasons other than ID and/or anticipated non-response to iron-supplementation (e.g. hemogobinopathy, bone marow disease, active cancer, unresolved active bleeding)
* Chronic liver disease (including active hepatitis) and/or screening alanine transaminase or aspartate transaminase above three times the upper limit of the normal range.
* Renal dialysis (previous, current, or planned within the next 6 months) or MDRD/CKD-EPI estimated glomerular filtration rate <15 mL/min.
* History of iron overload
* History of erythropoietin, i.v. or oral iron therapy, and blood transfusion in previous 3 months and/or such therapy planned within next 6 months
* Clinically apparent infection requiring antibiotic treatment
* Known hypersensitivity to iFCM or to any of its excipients
* Pregnancy
* Study subject participation in another TAVI related clinical study in which the primary endpoint includes mortality, hospitalization for heart failure and/or quality of life assessment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in Health-related Quality of Life (HRQOL) | The KCCQ-23 will be filled out pre-TAVI during an outpatient or inpatient geriatric visit, or at home and will be filled out again at week-24 post-TAVI during outpatient visit or at home.
  The primary endpoint is the change in HRQOL from baseline (pre-TAVI) to week-24 using the 23-item Kansas City Cardiomyopathy Questionnaire (KCCQ-23) which has been validated in patients undergoing TAVI.
Change in 6-Minute Walk Test (6-MWT) | 6-MWT is performed pre-TAVI during an outpatient or inpatient geriatric visit and will be measured again at week-24 post-TAVI during outpatient visit.
  The co-primary endpoint is change in exercise capacity from baseline (pre-TAVI) to week-24 using the 6-MWT, which is an established objective means of evaluation exercise capacity in the TAVI population.

SECONDARY OUTCOMES:
Cognitive function (MMSE) | Measured at week-24 post-TAVI
  Cognitive function using the Mini Mental State Examination (MMSE)
New York Heart Association (NYHA) functional class | Measured at week-24 post-TAVI
European Quality of Life-5 Dimensions 5 Level Utility Index (EQ-5D-5L-UI) and Visual Analog Scale (EQ-5D-VAS) | Measured at week-24 post-TAVI
  EQ5D comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels (no, slight, moderate, severe, and extreme problems) by which a unique health state per item is determined. These health states are converted into weighted health states (Utility Index or EQ-5D-5L-UI) by applying scores on which full health has a value of 1 and death a value of 0. The Visual Analog Scale (EQ-5D-VAS) is a self-reported score ranging from 0-100 with higher scores indicating better health.
Composite of cardiovascular mortality and heart failure hospitalizations | Measured at week-24 post-TAVI
All-cause mortality | Measured at week-24 post-TAVI
Favourable quality of life (QoL) | Measured at baseline (pre-TAVI) and week-24 post-TAVI
  Favourable QoL is defined as survival with a KCCQ-score ≥60 without KCCQ-decline >10 points from baseline to follow-up (week-24 post-TAVI)
Patient Global Assessment | Measured at week-24 post-TAVI

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands